CLINICAL TRIAL: NCT01941030
Title: Complete Lesion Assessment With ffR and IVUS TechnologY (CLARITY I)
Brief Title: Complete Lesion Assessment With ffR and IVUS TechnologY
Acronym: CLARITY I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLARITY I
Record Dates: First submitted 2013-03-11; First posted 2013-09-13 (Estimated); Results first posted 2019-01-24 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Peripheral Artery Disease; Critical Limb Ischemia
Keywords: Peripheral Artery Disease; Critical Limb Ischemia; Orbital Atherectomy; Balloon Angioplasty; Intravascular Ultrasound (IVUS); Fractional Flow Reserve (FFR)
MeSH Terms: conditions — Peripheral Arterial Disease; Chronic Limb-Threatening Ischemia | interventions — Angioplasty, Balloon

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Orbital Atherectomy System (Experimental): Orbital Atherectomy (OA) is performed prior to adjunctive Balloon Angioplasty (BA)
  Interventions: Device: Orbital Atherectomy System; Device: Balloon Angioplasty
- Balloon Angioplasty (Active Comparator): Balloon Angioplasty (BA) alone
  Interventions: Device: Balloon Angioplasty

INTERVENTIONS:
Device: Orbital Atherectomy System — Orbital atherectomy (OA) is performed prior to adjunctive balloon angioplasty (BA)
  Arms: Orbital Atherectomy System
Device: Balloon Angioplasty — Type of balloon selected is driven by preference of the operator.

SUMMARY:
CLARITY I is a pilot study to identify the clinically appropriate endpoint(s) of a larger, statistically powered pivotal trial for treatment of patients with Critical Limb Ischemia (CLI).

DETAILED DESCRIPTION:
This prospective, randomized, multi-center, post-market study of approximately 50 subjects randomized 1:1 to Orbital Atherectomy (OA) performed with Cardiovascular Systems, Inc.'s Orbital Atherectomy System (OAS) followed by adjunctive balloon angioplasty (BA) vs. BA alone for treatment of tibial vessel disease, defined as ≥ 50 % stenosis of the anterior tibial (AT), posterior tibial (PT), tibial peroneal trunk (TPT), or peroneal (PR) arteries by angiography. All subjects will have a corresponding wound being fed by the target vessel which will be assessed during the study. Subjects will be followed to one year.

ELIGIBILITY:
General Inclusion Criteria:

1. Subject's age ≥ 18 years.
2. Subject is an acceptable candidate for percutaneous intervention with the Sponsor's OAS and BA in accordance with their labeled indications and instructions for use.
3. Subject is willing and able to sign an approved informed consent form (ICF).
4. Subject is willing and able to attend follow-up and wound care visits.

General Exclusion Criteria:

1. Subject is pregnant or planning to become pregnant within the study period.
2. Subject is currently participating in an investigational drug or other device study that can clinically interfere with the endpoints of this trial.
3. Subject has a known sensitivity to contrast media and the sensitivity cannot be adequately pre-medicated.
4. Uncontrolled allergy to nitinol, stainless steel, or other stent materials.
5. Subject has known allergy to atherectomy lubricant components such as soybean oil, egg yolk phospholipids, glycerin or sodium hydroxide.
6. Subject has a history of bleeding diathesis or coagulopathy or will refuse blood transfusions.
7. Subject has been diagnosed with chronic renal failure or has a creatinine level > 2.5, unless on dialysis, prior to the index treatment.
8. Subject has evidence of intracranial or gastrointestinal bleeding within 90 days.
9. Subject has a history of trauma, fracture, major surgery (includes major amputation), or biopsy of a parenchymal organ within past 14 days, or patient has not healed from a previous medical intervention occurring more than 14 days.
10. Subject has a history of stroke or myocardial infarction (MI) within 90 days prior to enrollment in the study.
11. Subject has a planned major surgery (includes major amputation) scheduled within 60 days after treatment of the index limb.
12. Subject has a planned interventional treatment to address stenosis of the contralateral limb scheduled within 60 days after the index treatment.
13. Subject has a planned interventional treatment to address inflow stenosis of the ipsilateral limb scheduled within 60 days after the index treatment.
14. Inflow or bilateral PAD requiring treatment prior to enrollment was not successfully treated, defined as > 50% residual stenosis and/or occurrence of procedural angiographic complications, excluding dissection types A and B.
15. Subject has previously had their other limb treated as part of the study.

Angiographic Inclusion Criteria:

1. Target lesion(s) located in the anterior tibial (AT), posterior tibial (PT), tibial peroneal trunk (TPT) or peroneal (PR) arteries.
2. Target lesion has ≥ 50 % stenosis by angiography.
3. Subject has a corresponding wound being fed by the target vessel.

Angiographic Exclusion Criteria:

1. Target limb does not have any visual flow to the foot confirmed via distal selective angiography.
2. Thrombus is present or suspected in the target treatment vessel.
3. Target lesion is within a bypass graft or near a previously placed stent.
4. The guide wire cannot be passed across the target lesion.
5. Anterograde access of the lesion is not possible.
6. Subject has angiographic evidence of significant dissection at or near the treatment site.
7. Interventional treatment is intended for in-stent restenosis at the peripheral vascular site.
8. Subject's wound(s) involve multiple angiosomes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Dattilo, M.D., Principal Investigator — St. Francis Heart and Vascular Center
Locations (8):
- United States (8):
  - Arkansas Heart Clinic, Little Rock, Arkansas
  - Northside Hospital, Atlanta, Georgia
  - Midwest Cardiovascular Research Foundation, Davenport, Iowa
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Holy Name Medical Center, Teaneck, New Jersey
  - Rex Hospital, Raleigh, North Carolina
  - Mission Research Institute, New Braunfels, Texas
  - Sentara Vascular Specialists, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Started | 25 | 26
Completed | 12 | 13
Not Completed | 13 | 13
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 6 | 5
Not completed — Withdrawal by Subject | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Orbital Atherectomy System: Orbital Atherectomy (OA) is performed prior to adjunctive Balloon Angioplasty (BA) Orbital Atherectomy System: Orbital atherectomy (OA) is performed prior to adjunctive balloon angioplasty (BA) Balloon Angioplasty: Type of balloon selected is driven by preference of the operator.
- Balloon Angioplasty: Balloon Angioplasty (BA) alone Balloon Angioplasty: Type of balloon selected is driven by preference of the operator.
- Total: Total of all reporting groups
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.3 (11.3) | 69.4 (12.4) | 67.4 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 12 | 15
  Male | 22 | 14 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 3 | 9
  Not Hispanic or Latino | 19 | 23 | 42
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 8 | 16
  White | 17 | 18 | 35
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 26 | 51
Number of treated lesions [Number; unit: lesions] | 26 | 26 | 52

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Calcium Removal Out of Lumen Gain as Assessed by IVUS
Description: The post-treatment percentage of calcium removal out of lumen gain at the maximum calcium ablation site. A positive value equates to reduction in calcium out of the lumen gain.
Time Frame: Post-balloon angioplasty
Population: Not all subjects had reported IVUS data for each lesion pre- and post-treatment.
Measure: Median (Inter-Quartile Range); unit: percentage of lumen gain
Units Other Than Participants: lesions
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Number analyzed (Participants) | 25 | 26
Number analyzed (lesions) | 26 | 26
percentage of lumen gain | 25.0 [11.1 to 42.9] | 0.0 [0.0 to 6.7]
Statistical Analysis 1: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-balloon angioplasty reduction of calcium out of lumen gain; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.0220, Wilcoxon (Mann-Whitney); Data failed to meet the assumption for normality per the Shapiro-Wilk test

2. Primary Outcome: Change in Minimum Lumen Area Percent Stenosis as Assessed by IVUS
Description: The pre- (Pre-Tx) and post-treatment (Post-Tx) minimum lumen area percent stenosis. A positive value equates to a decrease in lumen area percent stenosis.
Time Frame: Pre-intervention, and post-balloon angioplasty
Population: Not all subjects had reported IVUS data for each lesion pre- and post-treatment.
Measure: Median (Inter-Quartile Range); unit: percent of minimum area stenosis
Units Other Than Participants: lesions
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Number analyzed (Participants) | 25 | 26
Number analyzed (lesions) | 26 | 26
percent of minimum area stenosis
  Pre-Tx, minimum area stenosis (%): number analyzed (lesions) | 17 | 21
  Pre-Tx, minimum area stenosis (%) | 43.8 [37.6 to 62.4] | 45.2 [34.5 to 58.5]
  Post-Tx, minimum area stenosis (%): number analyzed (lesions) | 19 | 20
  Post-Tx, minimum area stenosis (%) | 36.4 [29.0 to 51.5] | 31.5 [26.5 to 45.2]
Statistical Analysis 1: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-balloon angioplasty minimum lumen area stenosis; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.6228, t-test, 2 sided

3. Primary Outcome: Change in Plaque Area as Assessed by IVUS
Description: The pre- (Pre-Tx) and post-treatment (Post-Tx) plaque area. A positive value equates to a decrease in plaque area.
Time Frame: Pre-intervention, and post-balloon angioplasty
Population: Not all subjects had reported IVUS data for each lesion pre- and post-treatment.
Measure: Median (Inter-Quartile Range); unit: area (mm^3/mm)
Units Other Than Participants: lesions
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Number analyzed (Participants) | 25 | 26
Number analyzed (lesions) | 26 | 26
area (mm^3/mm)
  Pre-Tx, plaque area (mm^3/mm): number analyzed (lesions) | 19 | 22
  Pre-Tx, plaque area (mm^3/mm) | 6.5 [4.7 to 8.2] | 6.0 [4.9 to 6.5]
  Post-Tx, plaque area (mm^3/mm): number analyzed (lesions) | 19 | 21
  Post-Tx, plaque area (mm^3/mm) | 6.3 [4.4 to 10.0] | 6.0 [5.6 to 7.1]
Statistical Analysis 1: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-balloon angioplasty plaque area; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.4528, Wilcoxon (Mann-Whitney); Data failed to meet the assumption for normality per the Shapiro-Wilk test

4. Primary Outcome: Change in Dense Calcium Area as Assessed by IVUS
Description: The pre- (Pre-Tx) and post-treatment (Post-Tx) dense calcium area. A positive value equates to a decrease in dense calcium area.
Time Frame: Pre-intervention, and post-balloon angioplasty
Population: Not all subjects had reported IVUS data for each lesion pre- and post-treatment.
Measure: Median (Inter-Quartile Range); unit: area (mm^3/mm)
Units Other Than Participants: lesions
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Number analyzed (Participants) | 25 | 26
Number analyzed (lesions) | 26 | 26
area (mm^3/mm)
  Pre-Tx, dense calcium area (mm^3/mm): number analyzed (lesions) | 16 | 17
  Pre-Tx, dense calcium area (mm^3/mm) | 0.7 [0.2 to 1.5] | 1.0 [0.2 to 1.4]
  Post-Tx, dense calcium area (mm^3/mm): number analyzed (lesions) | 14 | 16
  Post-Tx, dense calcium area (mm^3/mm) | 0.4 [0.2 to 1.2] | 1.1 [0.2 to 1.7]
Statistical Analysis 1: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-balloon angioplasty dense calcium area; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.3573, Wilcoxon (Mann-Whitney); Data failed to meet the assumption for normality per the Shapiro-Wilk test

5. Primary Outcome: Change in Necrotic Core Area as Assessed by IVUS
Description: The pre- (Pre-Tx) and post-treatment (Post-Tx) necrotic core area. A positive value equates to a decrease necrotic core area.
Time Frame: Pre-intervention, and post-balloon angioplasty
Population: Not all subjects had reported IVUS data for each lesion pre- and post-treatment.
Measure: Median (Inter-Quartile Range); unit: area (mm^3/mm)
Units Other Than Participants: lesions
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Number analyzed (Participants) | 25 | 26
Number analyzed (lesions) | 26 | 26
area (mm^3/mm)
  Pre-Tx, necrotic core area (mm^3/mm): number analyzed (lesions) | 16 | 17
  Pre-Tx, necrotic core area (mm^3/mm) | 0.7 [0.4 to 1.2] | 0.9 [0.4 to 1.2]
  Post-Tx, necrotic core area (mm^3/mm): number analyzed (lesions) | 14 | 16
  Post-Tx, necrotic core area (mm^3/mm) | 0.8 [0.3 to 1.0] | 1.0 [0.5 to 1.1]
Statistical Analysis 1: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-balloon angioplasty necrotic core area; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.6073, Wilcoxon (Mann-Whitney); Data failed to meet the assumption for normality per the Shapiro-Wilk test

6. Primary Outcome: Change in Fibrous Plaque Area as Assessed by IVUS
Description: The pre- (Pre-Tx) and post-treatment (Post-Tx) fibrous plaque area. A positive value equates to a decrease in fibrous plaque area.
Time Frame: Pre-intervention, and post-balloon angioplasty
Population: Not all subjects had reported IVUS data for each lesion pre- and post-treatment.
Measure: Median (Inter-Quartile Range); unit: area (mm^3/mm)
Units Other Than Participants: lesions
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Number analyzed (Participants) | 25 | 26
Number analyzed (lesions) | 26 | 26
area (mm^3/mm)
  Pre-Tx, fibrous plaque area (mm^3/mm): number analyzed (lesions) | 16 | 17
  Pre-Tx, fibrous plaque area (mm^3/mm) | 1.7 [0.9 to 2.6] | 1.0 [0.6 to 2.0]
  Post-Tx, fibrous plaque area (mm^3/mm): number analyzed (lesions) | 14 | 16
  Post-Tx, fibrous plaque area (mm^3/mm) | 1.4 [0.9 to 3.3] | 0.9 [0.8 to 1.6]
Statistical Analysis 1: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-balloon angioplasty fibrous plaque area; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.2149, Wilcoxon (Mann-Whitney); Data failed to meet the assumption for normality per the Shapiro-Wilk test

7. Primary Outcome: Change in Fibrofatty Plaque Area as Assessed by IVUS
Description: The pre- (Pre-Tx) and post-treatment (Post-Tx) fibrofatty plaque area. A positive value equates to a decrease in fibrofatty plaque area.
Time Frame: Pre-intervention, and post-balloon angioplasty
Population: Not all subjects had reported IVUS data for each lesion pre- and post-treatment.
Measure: Median (Inter-Quartile Range); unit: area (mm^3/mm)
Units Other Than Participants: lesions
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Number analyzed (Participants) | 25 | 26
Number analyzed (lesions) | 26 | 26
area (mm^3/mm)
  Pre-Tx, fibrofatty plaque area (mm^3/mm): number analyzed (lesions) | 16 | 17
  Pre-Tx, fibrofatty plaque area (mm^3/mm) | 0.2 [0.1 to 0.7] | 0.1 [0.0 to 0.3]
  Post-Tx, fibrofatty plaque area (mm^3/mm): number analyzed (lesions) | 14 | 16
  Post-Tx, fibrofatty plaque area (mm^3/mm) | 0.2 [0.1 to 1.0] | 0.1 [0.0 to 0.1]
Statistical Analysis 1: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-balloon angioplasty fibrofatty plaque area; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.0579, Wilcoxon (Mann-Whitney); Data failed to meet the assumption for normality per the Shapiro-Wilk test

8. Secondary Outcome: Fractional Flow Reserve
Description: Fractional flow reserve (FFR) will be measured to assess hemodynamic function following each device procedure. During FFR, adenosine will be given through the femoral artery sheath or access catheter in two doses: 600 mcg and 1200 mcg. A higher FFR is presumed to correlate to better flow which may improve wound healing.
Time Frame: Post-orbital atherectomy (OA arm only) and post-balloon angioplasty (both arms)
Population: Some sites were exempt from performing FFR. Not all subjects had available FFR.
Measure: Mean (Standard Deviation); unit: Ratio (proximal/distal pressure)
Units Other Than Participants: lesions
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
Number analyzed (Participants) | 25 | 26
Number analyzed (lesions) | 26 | 26
Ratio (proximal/distal pressure)
  Post final OAS: FFR w/ 600 mcg adenosine: number analyzed (lesions) | 9 | 26
  Post final OAS: FFR w/ 600 mcg adenosine | 0.83 (0.14) | NA (NA) — Post final OAS value provided. OAS not used in Balloon Angioplasty arm.
  Post final OAS: FFR with 1200 mcg adenosine: number analyzed (lesions) | 9 | 26
  Post final OAS: FFR with 1200 mcg adenosine | 0.80 (0.12) | NA (NA) — Post final OAS value provided. OAS not used in Balloon Angioplasty arm.
  Post final balloon: FFR w/ 600 mcg adenosine: number analyzed (lesions) | 10 | 13
  Post final balloon: FFR w/ 600 mcg adenosine | 0.90 (0.13) | 0.75 (0.22)
  Post final balloon: FFR w/ 1200 mcg adenosine: number analyzed (lesions) | 10 | 13
  Post final balloon: FFR w/ 1200 mcg adenosine | 0.87 (0.10) | 0.76 (0.24)
Statistical Analysis 1: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-final balloon FFR value with 600 mcg adenosine; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.076, t-test, 2 sided
Statistical Analysis 2: Comparison: Orbital Atherectomy System vs Balloon Angioplasty; Null hypothesis: no difference in populations for post-final balloon FFR value with 1200 mcg adenosine; Test type: Other — No pre-specified hypothesis test or power calculation specified in protocol; p = 0.205, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: AEs were collected during the index-procedure through 12 months of follow-up.
Arm/Group | Orbital Atherectomy System | Balloon Angioplasty
All-Cause Mortality (participants affected / at risk) | 3/25 | 3/26
Serious Adverse Events (participants affected / at risk) | 22/25 | 17/26
Other Adverse Events (participants affected / at risk) | 4/25 | 8/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orbital Atherectomy System (N=25) | Balloon Angioplasty (N=26)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cellulitis, index limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Congestive Heart Failure (Cardiac disorders) | 2 (2) | 2 (3)
Coronary Artery disease, worsening (Cardiac disorders) | 1 (1) | 2 (2)
Deep Vein Thrombosis, upper arm (Vascular disorders) | 0 (0) | 1 (1)
Death, cardiac (Cardiac disorders) | 1 (1) | 0 (0)
Death, non-cardiac (General disorders) | 0 (0) | 2 (2)
Death, unknown cause (General disorders) | 2 (2) | 1 (1)
Dissection (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Distal embolization (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
GI bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hernia repair (Surgical and medical procedures) | 0 (0) | 1 (1)
Infection, other (Infections and infestations) | 0 (0) | 2 (2)
Major amputation, index limb, due to infected knee replacement (Surgical and medical procedures) | 1 (1) | 0 (0)
Major amputation, index limb due to gangrene (Surgical and medical procedures) | 2 (2) | 1 (1)
Major amputation, index limb due to osteomyelitis (Surgical and medical procedures) | 1 (1) | 0 (0)
Medication overdose (General disorders) | 0 (0) | 1 (1)
Medication side effect (General disorders) | 0 (0) | 1 (1)
Minor amputation - pre-planned, index limb (Surgical and medical procedures) | 2 (2) | 4 (4)
Minor amputation, index limb due to gangrene (Surgical and medical procedures) | 2 (2) | 2 (2)
Minor amputation, index limb due to osteomyelitis (Surgical and medical procedures) | 1 (1) | 1 (1)
Minor amputation, non-index limb due to gangrene (Surgical and medical procedures) | 1 (1) | 0 (0)
Minor amputation, non-index limb due to osteomyelitis (Surgical and medical procedures) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Osteomyelitis, index limb (Infections and infestations) | 0 (0) | 2 (2)
Osteomyelitis, non-index limb (Infections and infestations) | 0 (0) | 1 (1)
Other - Syncope (General disorders) | 1 (1) | 0 (0)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Recoil (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Revascularization - pre-planned, non-index limb (Surgical and medical procedures) | 1 (1) | 1 (1)
Revascularization, index limb (non-TVR) (Surgical and medical procedures) | 1 (1) | 3 (5)
Revascularization, index limb (TLR) (Surgical and medical procedures) | 3 (3) | 3 (3)
Revascularization, non-index limb (Surgical and medical procedures) | 4 (4) | 2 (6)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Worsening of index wound (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Orbital Atherectomy System (N=25) | Balloon Angioplasty (N=26)
Access site bleeding (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Dissection (Injury, poisoning and procedural complications) | 1 (1) | 5 (5)
Lower extremity edema (General disorders) | 0 (0) | 1 (1)
Pseudoaneurysm, access site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Slow flow (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 1 (1)
Vessel spasm (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
CLARITY I was a non-powered trial without a hypothesis test of a small number of patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less